CLINICAL TRIAL: NCT02244671
Title: Botulinum-assisted Orbital Fat Augmentation With PRP (Platelet-rich-plasma)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fox, Donald Munro, M.D., P.C. (Individual)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13.27
Record Dates: First submitted 2014-08-21; First posted 2014-09-19 (Estimated); Last update posted 2018-08-20 (Actual); Status verified 2018-08

CONDITIONS: Orbital Atrophy
MeSH Terms: interventions — CD36 Antigens; Botulinum Toxins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- fat, PRP, botulinum toxin (Experimental): Fat injection with platelet-rich-plasma (PRP) after immobilizing the extraocular muscles with botulinum toxin
  Interventions: Procedure: fat, PRP, botulinum toxin; Drug: botulinum toxin; Device: PRP

INTERVENTIONS:
Procedure: fat, PRP, botulinum toxin — fat injection with platelet-rich-plasma (PRP) after immobilizing the extraocular muscles with botulinum toxin
  Other Names: fat atrophy, absence of original eye, phthisis bulbi
Drug: botulinum toxin — botulinum toxin used to immobilize extra-ocular muscles prior to fat injection.
  Other Names: botulinum toxins
Device: PRP — autologous PRP is prepared with a dedicated centrifuge at the time of fat harvesting
  Other Names: platelet rich plasma

SUMMARY:
immobilization of yoked extra-ocular muscles in the anophthalmic orbit, in conjunction with platelet-rich-plasma, will improve integration of viable adipocytes injected into orbital fat

DETAILED DESCRIPTION:
Immobilization of tissue (graft, graft bed) is a prerequisite for tissue integration. Since yoked extra-ocular muscles continue to be stimulated by movements of the seeing eye after fat injection into the anophthalmic orbit, the use of botulinum toxin(s) can be used to prevent movement of the orbital tissue bed(s) and improve anchoring of injected fat. Platelet rich plasma may also improve fat cell anchoring by the action of fibrin on the adhesion process. This innovation builds on the results of IRB protocols 10.27 and 12.01 as registered with Clinical Trials.gov

ELIGIBILITY:
Inclusion Criteria:

* anophthalmic enophthalmos in subjects within a 50 mile radius of New York City, grade 0-1 anesthesia risk, ages 21-75

Exclusion Criteria:

* radiated orbits

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2014-01; Primary Completion 2018-01-03 (Actual); Study Completion 2018-01-03 (Actual)

PRIMARY OUTCOMES:
Orbital volume | one year
  Augmentation of orbital volume accessed with clinical photographs and non-contrast MRI

CONTACTS AND LOCATIONS:
Overall Officials: Donald M Fox, MD, Principal Investigator — New York Eye and Ear Infirmary
Locations (1):
- New York Eye and Ear Infirmary, New York, New York, United States

REFERENCES:
- See also: fat grafting — http://www.newyorkfami.com